CLINICAL TRIAL: NCT06923761
Title: A Modular, Multi-part, Multi-arm, Open-label, Phase I/II Study to Evaluate the Safety and Tolerability of GRWD5769 Alone and in Combination With Anticancer Treatments in Patients With Solid Malignancies
Brief Title: EMITT-1 (ERAP Mediated Immunopeptidome Targeting Trial - 1)
Acronym: EMITT-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grey Wolf Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GRWD5769-ST-01
Record Dates: First submitted 2025-03-27; First posted 2025-04-11 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Malignancy
Keywords: Oncology; ERAP 1; Solid tumors; TMB-H; NSCLC; Lung cancer; Cervical cancer; HCC - Hepatocellular Carcinoma; Liver cancer; Head and Neck Squamous Cell Carcinoma; SCCHN; Urothelial cancer; immuno oncology
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Hepatocellular; Liver Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Module 1 (GRWD5769 on its own as monotherapy) (Experimental)
  Interventions: Drug: Module 1 (GRWD5769 on its own as monotherapy)
- Module 2 (GRWD5769 in combination with cemiplimab, administered IV) (Experimental)
  Interventions: Drug: Module 2 (GRWD5769 in combination with cemiplimab, administered IV)

INTERVENTIONS:
Drug: Module 1 (GRWD5769 on its own as monotherapy) — Module 1 will initially be conducted in 4 study parts:
  Part A: Monotherapy dose escalation (where the safety of increasing doses of GRWD5769 will initially be assessed in a small group of patients, overseen by a safety review committee)
  Part B: (Optional) Monotherapy dose expansion part (to look at the effect of GRWD5769 on the body, and of the body on GRWD5769, at particular dose levels to include evaluation of biopsies of tumour tissue)
  Part C: (Optional) Intra-patient dose escalation (where a patient may receive three different GRWD5769 doses so that blood levels at each dose can be measured in an individual)
  Part D: Monotherapy dose expansion group(s) (where a dose of GRWD5769 may be chosen to be evaluated in specific types of cancer)
  Arms: Module 1 (GRWD5769 on its own as monotherapy)
Drug: Module 2 (GRWD5769 in combination with cemiplimab, administered IV) — Module 2 will initially be conducted as 3 study parts, similar to those above, but looking at GRWD5769 when given in combination with cemiplimab:
  Part A: Combination therapy dose escalation (like Module 1 Part A)
  Part B: (Optional) Combination therapy dose expansion part (like Module 1 Part B)
  Part C: Combination therapy dose expansion group(s) (where a dose of GRWD5769 given with cemiplimab will be evaluated in specific types of cancer)
  Part D: Randomised dose optimisation, combination therapy (where 3 doses of GRWD5769 given with cemiplimab will be evaluated in specific types of cancer)
  Arms: Module 2 (GRWD5769 in combination with cemiplimab, administered IV)

SUMMARY:
This is a Phase I/II, open-label, first-in human study of GRWD5769 alone, and in combination with another anti-cancer agent in advanced solid cancers.

DETAILED DESCRIPTION:
GRWD5769 is as a potential new treatment for advanced or metastatic solid malignancies. GRWD5769 works by stopping an enzyme in the body, called endoplasmic reticulum aminopeptidase 1 (ERAP1), from working. ERAP1 is part of how the body recognizes the presence of a cancer tumour and helps trigger the immune system to fight the cancer. However, in patients with cancer, the immune system cells can become exhausted and no longer work effectively. By blocking ERAP1 it makes the tumour look different to the immune system and so the immune system starts fighting the cancer again. GRWD5769 has the potential of producing clinically meaningful improvements in monotherapy and in combination with therapy like cemiplimab (Libtayo®) by enhancing the antitumour immune response.

Who can participate? Patients with advanced or metastatic solid malignancy aged 18 years or older.

What does the study involve? This study consists of Module 1 (Parts A to D), which will look at the effects of GRWD5769 when given alone and Module 2 (Parts A to D) which will look at the effects of GRWD5769 when given in combination with another anticancer drug called Libtayo® (cemiplimab).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent.
2. Male or female, ≥ 18 years of age.
3. An ECOG performance status of 0 or 1.
4. Willing to permit access to stored historical tumour tissue and prior tumour radiological assessments and tumour biomarker data (if available).
5. Able to take oral medications and be willing to record daily adherence to the study drug.
6. Female participants must be of non-child-bearing potential, or, if of childbearing potential must have a negative pregnancy test (as required by protocol), must use a highly effective method of contraception combined with a condom and not donate ova (for the protocol specified period of time).
7. Male participants must use a condom and their female participant must also use a highly effective method of contraception (for the protocol specified period of time), if engaging in sexual intercourse with a female partner who could become pregnant and not donate sperm.
8. Estimated life expectancy of at least 3 months, in the opinion of the PI.
9. Willing and able to comply with all scheduled visits, treatment plans, laboratory tests, and other study procedures.
10. Participant has measurable disease per RECIST 1.1/iRECIST
11. Participant has cytologically or histologically confirmed locally advanced or metastatic solid malignancy for which no further standard of care (SoC) therapy is available (or no SoC therapy exists), or who have been offered and declined SoC therapy, or are intolerant of SoC therapy.

    Module 1 (Part B) and Module 2 (Part B) Only
12. Participant has at least one tumour lesion amenable to serial biopsies and is willing to provide consent for biopsies and has measurable disease per RECIST 1.1/iRECIST, excluding the lesion(s) identified for biopsy.

    Module 2 (Part C and Part D)

    Cohort 1 (Cervical)
13. Participants with histologically confirmed persistent, recurrent or metastatic cervical cancer who are not amenable to curative therapy.
14. Participants should have received at least 3 months first line anti-PD(L)-1 therapy (± bevacizumab, chemotherapy, ADC or other immunotherapy e.g. anti-CTLA-4) and this should have included at least a 10-week period without progression.
15. Participants may enrol in the study immediately following progression on the first line CPI or may have received 1 further line of systemic cancer therapy after progression on CPI.

    Cohort 2 (Hepatocellular Carcinoma)
16. Participants with histologically confirmed hepatocellular carcinoma who are not amenable to curative therapy and ineligible for loco-regional therapy.
17. Participants should have received at least 3 months first line anti-PD(L)-1 containing therapy and this should have included at least a 10-week period without progression per Investigator assessment.
18. Participants may enrol in the study immediately following progression on the first line CPI or may have received 1 further line of systemic cancer therapy after progression on CPI.
19. Participant has Child-Pugh score class A liver function.

    Cohort 3 (Moderate to High TMB)
20. Participants with cytologically or histologically confirmed advanced, recurrent or metastatic disease, which is not amenable to curative therapy, in up to 5 types of solid tumour with moderate to high median TMB (NSCLC, urothelial, SCCHN, gastric/gastro-oesophageal adenocarcinoma, oesophageal SCC).
21. Participants should have received at least ≥ 3 months first line anti-PD(L)-1 (± chemotherapy, ADC, pemetrexed or other immunotherapy e.g. anti-CTLA-4) and this should have included at least a 10-week period without progression.
22. Participants may enrol in the study immediately following progression on the first line CPI or may have received 1 further line of systemic cancer therapy after progression on CPI.

    Module 2 Part D only (pMMR/MSS-CRC)
23. Participants with histologically confirmed unresectable pMMR/MSS-CRC, without current or prior liver metastases
24. Participants should have received at least one line of therapy in the advanced/metastatic setting and should have received therapies according to local standard practice, unless ineligible or intolerant to the treatment
25. Participants may not have received more than 2 lines of cytotoxic chemotherapy

Exclusion Criteria:

1. Prior therapy with an ERAP1 inhibitor.
2. Any other malignancy within the past 3 years, with the exception of cervical intraepithelial neoplasia and nonmelanoma skin cancer.
3. Any unresolved toxicity (except alopecia) from prior therapy of ≥ CTCAE Grade 1. Participants with Grade 2 toxicity that is not clinically significant (e.g., alopecia, vitiligo), or that is deemed stable or irreversible (e.g., peripheral neuropathy) can be enrolled.
4. Active or documented history of autoimmune disease (within 2 years) requiring systemic immunosuppressive therapy, or participant is immunocompromised for any other reason (as determined by the Investigator).
5. Spinal cord compression or brain metastases, unless asymptomatic, stable, and not requiring steroids for at least 4 weeks (if stable and requiring no intervention, the participant can be enrolled in the study).
6. Uncontrolled seizures.
7. Active infection requiring therapy within 14 days prior to the day of first dose of IMP.
8. Severe or uncontrolled medical condition (e.g., severe chronic obstructive pulmonary disease, severe Parkinson's disease, active inflammatory bowel disease) or psychiatric condition.
9. Active bleeding diatheses.
10. Participant has received an organ transplant.
11. Known active hepatitis B, hepatitis C, or human immunodeficiency virus infection (HIV).
12. Participant is breastfeeding or pregnant.
13. Receipt of licenced or unlicenced cytotoxic, noncytotoxic or small molecule treatment for the malignancy within 28 days or 5 half-lives, whichever is shorter prior to the day of first dose of IMP.
14. Receipt of oral corticosteroids (at a dose > 10 mg prednisone/day or equivalent) within 14 days (except for subjects receiving corticosteroids for adrenal insufficiency).
15. Receipt of St John's Wort or of another concomitant medication, herbal supplement, or food that is a strong inhibitor or inducer of CYP3A4 enzymes within 14 days.
16. Receipt of a blood transfusion (blood or blood products) within 7 days.
17. Impaired hepatic or renal function.
18. Liver function deteriorating in a manner that would likely make the participant ineligible per protocol specified requirements.
19. Other evidence of impaired hepatic synthesis function.
20. Inadequate bone marrow reserve or organ function.
21. Any prior history of persistent (> 4 weeks) severe pancytopenia due to previous therapy rather than to disease (ANC < 0.5 × 10^9/L or platelets < 50 x 10^9/L).
22. Cardiac dysfunction or other clinically significant cardiac pathology likely to impair the participants ability to participate in the study.
23. Mean QTcF > 450 ms for males or > 470 ms for females.
24. Any clinically important abnormalities in rhythm, conduction, or morphology on resting ECG. Controlled atrial fibrillation is permitted.
25. Any factor that in the Investigator's opinion increases the risk of QTc prolongation or arrythmic events.
26. In the opinion of the Investigator, unlikely to comply with study procedures, restrictions, or requirements.
27. A history of haemolytic anaemia or marrow aplasia.
28. Has received a live-virus vaccination within 28 days. Note: seasonal flu or COVID vaccines that do not contain live virus are permitted.
29. History of Grade 3 or 4 pneumonitis or interstitial lung disease within the last 5 years, or other clinically significant pulmonary pathology likely to impair ability to participate in the study.

    Module 2 all Parts and Module 1A Crossover Participants Only
30. Has discontinued a prior checkpoint inhibitor due to toxicity.
31. Hypersensitivity to cemiplimab or any of its excipients, or contraindicated to cemiplimab per approved local labelling.
32. Has experienced ≥ Grade 2 immune-mediated AE on this study (applies to crossover participants only).

    Module 2 Part D only - pMMR/MSS CRC dose optimisation cohort
33. Participants with unresectable pMMR/MSS CRC may not have purely peritoneal disease
34. Participants with unresectable pMMR/MSS CRC may not have had prior CPI / immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-21 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of treatment emergent and treatment related AEs | From first dose to 30 days after last dose of GRWD5769 for Module 1 and 90 days after last dose of cemiplimab for Module 2 Parts A-C.
  Incidence of treatment emergent and treatment related AEs assessed from start of study drug to 30 days post last dose of GRWD5769 (Module 1) or to 90 days post last dose of cemiplimab (Module 2 Parts A-C).
Incidence of Dose limiting toxicities (DLT) | End of cycle 1 (each cycle is 21 days)
  Incidence of Dose limiting toxicities (DLT) during the DLT period which commences Cycle 0 Day 1 and continues to 21 days after Cycle 1 Day 1
Comparative efficacy (for Module 2D only) | From baseline to week 16
  Comparative efficacy will be evaluated or assessed using the change in dimension over time of RECIST Target Lesions from baseline and on-study scans recorded at weeks 8 and 16

SECONDARY OUTCOMES:
GRWD5769 Plasma PK Trough concentration | Up to approximately 1 year
Objective response rate (ORR) | Up to approximately 1 year
  Preliminary efficacy of GRWD5769 will be assessed by:
  Tumour response (ORR) by RECIST 1.1 or iRECIST as determined by CT/MRI scans performed every 8 weeks until participant disease progression or withdrawal.
Disease specific tumour markers | Up to approximately 1 year
  Changes in any applicable disease-specific tumour markers assessed pre-treatment, Day 1 of each cycle from Cycle 2 onwards, at each 6-weekly safety extension visit, at the end of study visit and at follow up visit 30 days post last dose of GRWD5769.
GRWD5769 Plasma PK Cmax | Up to approximately 1 year
  Cmax = Maximum observed concentration
GRWD5769 Plasma PK Tmax | Up to approximately 1 year
  Tmax = Time to maximum observed concentration
GRWD5769 Plasma PK AUC0-t | Up to approximately 1 year
  AUC0-t = Area under the concentration-time curve
GRWD5769 Plasma PK Half-life | Up to approximately 1 year
GRWD5769 Plasma PK Oral Clearance | Up to approximately 1 year
GRWD5769 Plasma PK Vss/F | Up to approximately 1 year
  Vss/F = Absorption-dependent apparent volume of distribution in steady state
Disease Control Rate (DCR) | Up to approximately 1 year
  Preliminary efficacy of GRWD5769 will be assessed by:
  Tumour response (DCR) by RECIST 1.1 or iRECIST as determined by CT/MRI scans performed every 8 weeks until participant disease progression or withdrawal.
Stable Disease Rate (SDR) | Up to approximately 1 year
  Preliminary efficacy of GRWD5769 will be assessed by:
  Tumour response (SDR) by RECIST 1.1 or iRECIST as determined by CT/MRI scans performed every 8 weeks until participant disease progression or withdrawal.
Time To Response (TTR) | Up to approximately 1 year
  Preliminary efficacy of GRWD5769 will be assessed by:
  Tumour response (TTR) by RECIST 1.1 or iRECIST as determined by CT/MRI scans performed every 8 weeks until participant disease progression or withdrawal.
Duration Of Response (DOR) | Up to approximately 1 year
  Preliminary efficacy of GRWD5769 will be assessed by:
  Tumour response (DOR) by RECIST 1.1 or iRECIST as determined by CT/MRI scans performed every 8 weeks until participant disease progression or withdrawal.
Progression - Free Survival (PFS) | Up to approximately 1 year
  Preliminary efficacy of GRWD5769 will be assessed by:
  Tumour response (PFS) by RECIST 1.1 or iRECIST as determined by CT/MRI scans performed every 8 weeks until participant disease progression or withdrawal.
Number of treatment emergent and treatment related AEs (for Module 2D only) | 90 days after last dose of cemiplimab
  Incidence of treatment emergent and treatment related AEs assessed from start of study drug to 90 days post last dose of cemiplimab (for Module 2D only).
Incidence of Dose limiting toxicities (DLT) (for Module 2D only) | End of cycle 1 (each cycle is 21 days)
  Incidence of Dose limiting toxicities (DLT) during the DLT period which commences Cycle 0 Day 1 and continues to 21 days after Cycle 1 Day 1
Overall Survival | Up to approximately 1 year
  Preliminary efficacy of GRWD5769 will be assessed by:
  Overall survival assessed from start of study drug until participant withdrawal or death (for Module 2C and 2D only).

CONTACTS AND LOCATIONS:
Locations (29):
- Australia (8):
  - GenesisCare Research, Adelaide
  - Southern Oncology Clinical Research Unit (SOCRU), Bedford Park
  - Blacktown Hospital, Blacktown
  - Kinghorn Cancer Centre (KCC), Darlinghurst
  - Austin Health, Heidelberg
  - Alfred Health, Melbourne
  - Mater Research, South Brisbane
  - Cancer Care Wollongong, Wollongong
- France (7):
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre Eugène Marquis, Rennes
  - Institut de Cancérologie de l'Ouest (ICO), Saint-Herblain
  - ICANS - Institut de Cancérologie Strasbourg, Strasbourg
  - IUCT Oncopole - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Spain (8):
  - Hospital Universitario Vall d'Hebrón (VHIO), Barcelona
  - START Barcelona - Hospital HM Nou Delfos, Barcelona
  - Clinica Universitaria de Navarra Madrid, Madrid
  - START Madrid - Centro Integral Oncológico Clara Campal (HM CIOCC), Madrid
  - START Madrid - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Clinica Universitaria de Navarra Pamplona, Pamplona
  - INCLIVA-Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (6):
  - Western General Hospital, Edinburgh
  - Clatterbridge Cancer Centre, Liverpool
  - Hammersmith Hospitals NHS Trust, London
  - Royal Free Hospital, London
  - Christie NHS Foundation Trust, Manchester
  - Newcastle Upon Tyne Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: No
IPD may not be shared for this Phase 1 study, or the IPD plan may be updated at a later point.